CLINICAL TRIAL: NCT06587724
Title: Investigation of the Validity, Reliability, and Responsiveness of the BETY-Biopsychosocial Questionnaire in Individuals Diagnosed with Myositis
Brief Title: Investigation of the Validity, Reliability, and Responsiveness of the BETY-BQ in Myositis
Acronym: BETY-BQ
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: SBA 24/533
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myositis
Keywords: myositis; biopsychosocial model; validity and reliability; BETY-BQ; muscle strenght; pain
MeSH Terms: conditions — Myositis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire study — Questionnaire application
  Other Names: BETY-Biopsychosocial Questionnaire

SUMMARY:
Individuals diagnosed with myositis have skin, joint, and visceral organ involvement together with proximal muscle weakness, impaired physical function, sexual function, and quality of life also affect individuals psychosocially. Increased anxiety-depression-anxiety problems are observed in individuals, and many factors contributing to these conditions are reported. Therefore, while holistic evaluation of individuals, including these factors, gains importance, more information on how the quality of life changes during the disease is required. There is a need for tools to evaluate these characteristics in individuals disease management and treatment process.

The cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı-BETY) is an innovative exercise model based on physical exercise and an example of a biopsychosocial approach developed in patients with rheumatism. The BETY-Biopsychosocial Questionnaire (BETY-BQ) was created by repeated statistics of the improvement characteristics reported by individuals who participated in BETY sessions for many years. The BETY-BQ holistically evaluates many biopsychosocial characteristics of the individual, such as pain, coping skills, functionality, mood, sociability, sexuality, and sleep. Therefore, there is a need for scales that holistically evaluate the symptoms mentioned in myositis disease. Since the BETY-BQ can assess biopsychosocial characteristics quickly and its structure was created with the feedback of individuals with chronic disease, it aimed to examine its validation in this disease group.

This study, which the investigators planned to contribute to this field, aims to investigate BETY-BQ^s validity, reliability, and responsiveness in individuals diagnosed with myositis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myositis
* To be over 18 years old
* Consent of the participant

Exclusion Criteria:

* Uncontrolled/other clinically significant disease (chronic obstructive pulmonary disease, congestive heart failure, endocrine system diseases, neurological, psychological diseases, etc.) individuals with a diagnosis,
* Pregnant individuals,
* Individuals with malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire | Three months
  The biopsychosocial status of the individual is assessed with questions about pain, functionality, mood, sociability, sexuality, and sleep status. Each question consists of 30 items scored between 0-120 as '0 (never), 1 (yes rarely), 2 (yes sometimes), 3 (yes often), 4 (yes always)'. A high score indicates poor biopsychosocial status

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale | Three months
  It consists of 14 items, 7 of which assess anxiety, and the other 7 determine depression. Each item is scored between 0-3, and the total is scored between 0-21. High scores indicate poor anxiety and depression levels.
Myositis Disease Activity Assessment Tool (MDAAT) | Three months
  The Myositis Disease Activity Assessment Tool (MDAAT) is a tool that assesses the disease activity of non-muscle organ systems and muscles in patients with myositis. The MDAAT combined tool includes the Myositis Disease Activity Assessment VAS (MYOACT) and the Myositis Activities Index for Therapeutic Purposes (MITAX). MYOACT is a series of physician judgments of disease activity in various organ systems using a VAS to assess the severity of disease activity. MITAX indicates disease damage from myositis, in the physician's opinion. For MYOACT, each organ system receives a score of 0-10, and the six non-muscular organ systems are summed to obtain an extra-muscular score of 0-60 or a total score including the muscular system ranging from 0-60. For MITAX, each question is scored 0 = not available; 1 = improvement; 2 = same; 3 = worse; 4 = new. The organ system scores are summed to obtain a total MITAX score of 0-63 or 0-54 if the muscular system is excluded.
Health Assessment Questionnaire | Three months
  The Health Assessment Questionnaire evaluates the functionality of the individual using eight parameters and 20 items. The parameters are classified as dressing, standing, eating, walking, hygiene, reaching, grasping, and other activities. Each item is scored as 0 (without any difficulty), 1 (with some difficulty), 2 (with a lot of difficulty), and 3 (unable to do at all). The total score is between 0-3, with a high score indicating low functionality.
Dermatology Life Quality Index | Three months
  Ten questions assess the quality of life-related to dermatological findings. The first and second questions are about symptoms and feelings, the third and fourth questions are about daily activities, the fifth and sixth questions are about leisure time activities, the seventh question is about work and school, the eighth and ninth questions are about interpersonal relationships and the tenth question is about treatment. The items are scored as 3 (quite a lot), 2 (very much), 1 (slightly), 0 (not at all), 0 (not relevant) between 0-30. A high score indicates a decrease in quality of life.
Hand Dynamometer | Three months
  Muscle strength will be measured with a hand dynamometer (Lafayette Instrument®, Lafayette, IN) routinely used in the rheumatological rehabilitation unit. The dynamometer allows maximal isometric strength to be measured objectively and reliably using a standardized protocol. High values indicate a high strength value. In our study, deltoid, biceps, wrist extensors, quadriceps, gluteus maximus, gluteus medius, ankle dorsiflexion, and neck flexors isometric muscle strength values will be measured with a hand dynamometer in the appropriate evaluation position for each muscle. For each position, three measurements (3 seconds of contraction, 30 seconds of rest) will be made, and mean values will be calculated.
Timed Up and Go Test | Three months
  The balance status of the individual is evaluated by getting up from a back-supported chair and walking 3 meters at a normal walking speed and returning to the chair and the time of sitting on the chair is measured and recorded in seconds.
30 Seconds Sit to Stand Sest | Three months
  To evaluate lower extremity strength, the individual stands upright on a chair with his/her arms crossed on his/her chest and then sits down again. The individual is asked to repeat at his/her own pace for 30 seconds. The score of this assessment test is the number of times the individual stands up fully from a sitting position with arms crossed within 30 seconds.
10-Metre Walk Test | Three months
  The individual is asked to walk quickly without running on a 10-metre path. It is recorded in seconds in the evaluation made with three repetitions.
Short Form-36 | Three months
  Quality of life is a 36-item generic scale that assesses the quality of life with eight parameters (physical functioning, social functioning, role limitations due to physical complaints, role limitations due to emotional problems, mental health, energy-vitality, bodily pain (BP), general health perception), each parameter is scored between 0-100. A high score indicates a good quality of life.
Visual Analogue Scale | Three months
  The individual diagnosed with myositis will asked to show the pain, fatigue, and disease activity status in the last week on a 10 cm long Visual Analogue Scale (VAS). A high score shows worse pain, fatigue, and disease activity status.
Manual Muscle Test-8 | Three months
  The Manual Muscle Test-8 (MMT-8) is one of the most popular instruments for measuring muscle strength. It is a shorter version of the original instrument in which the individual^s eight dominant proximal, distal, and axial muscle groups are tested unilaterally. Each muscle group examined is scored from 0-10 (0 = extreme weakness and 10 = normal strength) depending on how much it can move against gravity or pressure applied by the examiner.
Stair Climb Test | Three months
  To measure the individual^s lower extremity strength and dynamic balance, the time to ascend and descend a 10-step staircase with a handrail in the range of 16-20 cm as fast as possible is recorded in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will not be shared to protect the data of individuals